CLINICAL TRIAL: NCT03289871
Title: Clinical Evaluation of the Efficacy of a Medical Device in Treatment of Toenail Onychomycosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oystershell NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14E0752
Record Dates: First submitted 2016-05-03; First posted 2017-09-21 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2016-05

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Excilor (Experimental): 2 applications per day for 6 months
  Interventions: Device: Excilor
- Loceryl 5% (Active Comparator): 1 application per week for 6 months
  Interventions: Drug: Loceryl 5%

INTERVENTIONS:
Device: Excilor
  Arms: Excilor
Drug: Loceryl 5%
  Arms: Loceryl 5%

SUMMARY:
This study evaluates the effect of the medical device "Excilor® Fungal Nail Infection" in the treatment of toenail onychomycosis. Half of the participants will receive the tested product and the other half will receive a comparator (Amorolfin 5%). Patients will be followed during 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject having given her/his informed, written consent,
* Subject cooperative and aware of the modalities of use and the necessity and duration of the controls so that perfect adhesion to the protocol can be expected.
* Subject being psychologically able to understand information and to give their/his/her consent.
* Age: more than 18 years.
* Subject with superficial onychomycosis on at least one great toenail or light to moderate disto-lateral onychomycosis (without matrix involvement and involvement <2/3 of the tablet).
* Subject with positive results of KOH staining.
* Subject having stopped any systemic antifungal treatment since at least 6 months before inclusion and/or any topical antifungal treatment since at least 3 months before inclusion.
* Female subjects of childbearing potential should use an accepted contraceptive regimen since at least 12 weeks before the beginning of the study, during all the study and at least 1 month after the study end.

Exclusion Criteria:

* Subject considered by the Investigator likely to be non-compliant with the protocol.
* Patient enrolled in another clinical trial during the test period.
* Woman being pregnant, nursing or planning a pregnancy during the course of this study.
* Subject having a known allergy to one of the constituents of the tested products.
* Patient suffering from serious or progressive diseases (to investigator's discretion), such as diabetes, peripheral circulatory disease, HIV, psoriasis, lichen planus, immunosuppressive pathology….
* Subject with cutaneous pathology on studied zone (other than onychomycosis like angioma, dermatitis…).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
At the end of the study (day 168), evolution of the percentage of healthy surface versus baseline, was evaluated by a blinded investigator. Comparison with the comparator product. | After 168 days of treatment
  Percentage healthy surface was assessed using digital image analysis. Briefly, two macro-photographs (top and front) were made of the great toenail, placed beside a piece of graph paper to allow determination of the exact size of the nail during analysis (contour tracing). Consequently, all pictures were digitalised and recorded on the computer. Image analysis of the top picture was performed with Adobe Photoshop software. For each photograph, a blinded dermatologist traced the healthy surface.

SECONDARY OUTCOMES:
At different time points, evolution of the percentage of healthy surface versus baseline, was evaluated by a blinded investigator. Comparison with the comparator product. | After 14, 28, 56 and 112 days of treatment
  Percentage healthy surface was assessed using digital image analysis. Briefly, two macro-photographs (top and front) were made of the great toenail, placed beside a piece of graph paper to allow determination of the exact size of the nail during analysis (contour tracing). Consequently, all pictures were digitalised and recorded on the computer. Image analysis of the top picture was performed with Adobe Photoshop software. For each photograph, a blinded dermatologist traced the healthy surface.
Evaluation of the clinical efficacy assessed by the investigator with structured scales. Comparison with the comparator product. | On Day 0, Day 14, Day 28, Day 56, Day 112 and Day 168
  Onycholysis, nail dystrophy, nail discoloration and nail thickening were assessed using the following scores:
  0 = none, 1 = very slight, 2 = slight, 3 =moderate, and 4 = severe.
Evaluation of the microbiological efficacy of the product assessed by fungal culture and comparison with the comparator product. | On baseline (day zero) and day 168
Evaluation of the product tolerance, assessed by the investigator by clinical evaluation and subject interrogatory with a score from 0 (bad tolerance) to 3 (very good tolerance). | After 14, 28, 56 and 112 days of treatment
Evaluation of the quality of life of the subjects thanks to the questionnaire NailQoL . Comparison with the comparator product. | On Day 0, Day 14, Day 28, Day 56, Day 112 and Day 168
Subjective evaluation by subjects by completing the subjective evaluation questionnaire at each visit. | On Day 0, Day 14, Day 28, Day 56, Day 112 and Day 168

CONTACTS AND LOCATIONS:
Overall Officials: Nejib Doss, MD, Principal Investigator — Principal Instruction military hospital of Tunis
Locations (2):
- Tunisia (2):
  - Hospital Habib Thameur, Tunis
  - Principal instruction military hospital, Tunis